CLINICAL TRIAL: NCT02436330
Title: Exergaming for Health: Impact of a Community-Based Active Video Gaming Curriculum in Pediatric Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Amy Christison, M.D., Associate Professor of Pediatrics, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 209418
Record Dates: First submitted 2015-04-20; First posted 2015-05-06 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Pediatric Obesity
Keywords: Exergaming, Weight management
MeSH Terms: conditions — Pediatric Obesity | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exergaming and Didactic health teaching (Experimental): Participation of child and parent/guardian in 6 months of weight management programming consisting of exergaming combined with didactic teaching.
  Interventions: Behavioral: Exergaming; Behavioral: Didactic health teaching
- Didactic health teaching (Active Comparator): Participation of child and parent/guardian in 6 months of weight management programming consisting only of didactic teaching.
  Interventions: Behavioral: Didactic health teaching

INTERVENTIONS:
Behavioral: Exergaming — 6 months of weight management programming consisting of 10 weekly sessions:1 hour of session was spent "exergaming", which included active video game play and traditional group exercises. Some examples include: Dance, Dance, Revolution, Exerbike, Treadwall, Yoga, Spin class, etc.
  Arms: Exergaming and Didactic health teaching
Behavioral: Didactic health teaching — 6 months of weight management programming consisting of 10 weekly 1-hour sessions of didactic classes teaching behavioral and dietary curricula. Followed by monthly 1 hour didactic health teaching sessions for the remainder of the 6 month period.

SUMMARY:
Evaluation of the effectiveness of Exergaming for Health, a community-based multifaceted weight management program in a randomized controlled trial (RCT). Primary objective: to assess impact of the program on BMI z-scores. Secondary objectives: to measure impact on cardiovascular fitness, self-worth, sedentary screen time, and the influence of exergaming component on attendance and participation.

DETAILED DESCRIPTION:
Eighty-four overweight pediatric subjects will be enrolled sequentially and randomized 2:1 in experimental and control groups for six months of weight management programming. The experimental group and their parents/guardians will participate in ten weekly 2-hour sessions, comprised of 1 hour of exergaming or exergaming combined with traditional exercise and 1 hour of didactic classes focusing on nutrition and psychosocial behaviors related to weight management. Following these 10 weeks, they will attend monthly 1-hour maintenance didactic classes. The control group and their parents/guardians will participate only in the didactic portion of the curricula for the same duration of time, 10 weeks, followed by monthly maintenance classes for the remainder of the 6 month period. The control group will then be offered participation in the Exergaming for Health program upon study completion.

Comparisons between the two groups will be obtained through changes in the measurements of weight, height, BMI z-scores, shuttle run times, and responses to questionnaires about screen time, self-perception, and nutrition. Measurements of both groups will be obtained at baseline and 6 months and another set of measurements will be obtained on the experimental group at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Child with BMI greater than or equal to 85th percentile.
* English speaking
* Approval by Primary Care Doctor

Exclusion Criteria:

* Participants with medical, developmental or psychiatric diagnoses which preclude participation in both the physical activity and classroom portions of the curriculum.
* Participants who are taking medications that positively or negatively affect weight.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy L. Christison, MD, Principal Investigator — University of Illinois College of Medicine at Peoria

REFERENCES:
- [Background] Sacher PM, Kolotourou M, Chadwick PM, Cole TJ, Lawson MS, Lucas A, Singhal A. Randomized controlled trial of the MEND program: a family-based community intervention for childhood obesity. Obesity (Silver Spring). 2010 Feb;18 Suppl 1:S62-8. doi: 10.1038/oby.2009.433. PMID 20107463
- [Background] Vandewater EA, Shim MS, Caplovitz AG. Linking obesity and activity level with children's television and video game use. J Adolesc. 2004 Feb;27(1):71-85. doi: 10.1016/j.adolescence.2003.10.003. PMID 15013261
- [Background] Gortmaker SL, Cheung LW, Peterson KE, Chomitz G, Cradle JH, Dart H, Fox MK, Bullock RB, Sobol AM, Colditz G, Field AE, Laird N. Impact of a school-based interdisciplinary intervention on diet and physical activity among urban primary school children: eat well and keep moving. Arch Pediatr Adolesc Med. 1999 Sep;153(9):975-83. doi: 10.1001/archpedi.153.9.975. PMID 10482216
- [Background] Robinson TN. Reducing children's television viewing to prevent obesity: a randomized controlled trial. JAMA. 1999 Oct 27;282(16):1561-7. doi: 10.1001/jama.282.16.1561. PMID 10546696
- [Background] Daley AJ. Can exergaming contribute to improving physical activity levels and health outcomes in children? Pediatrics. 2009 Aug;124(2):763-71. doi: 10.1542/peds.2008-2357. Epub 2009 Jul 13. PMID 19596728
- [Background] Lanningham-Foster L, Jensen TB, Foster RC, Redmond AB, Walker BA, Heinz D, Levine JA. Energy expenditure of sedentary screen time compared with active screen time for children. Pediatrics. 2006 Dec;118(6):e1831-5. doi: 10.1542/peds.2006-1087. PMID 17142504
- [Background] Ridley K, Olds T. Video center games: Energy cost and children's behaviors. Pediatric Exercise Science. 2001;13:413-421.
- [Background] Unnithan VB, Houser W, Fernhall B. Evaluation of the energy cost of playing a dance simulation video game in overweight and non-overweight children and adolescents. Int J Sports Med. 2006 Oct;27(10):804-9. doi: 10.1055/s-2005-872964. PMID 17006803
- [Background] Mellecker RR, McManus AM. Energy expenditure and cardiovascular responses to seated and active gaming in children. Arch Pediatr Adolesc Med. 2008 Sep;162(9):886-91. doi: 10.1001/archpedi.162.9.886. PMID 18762609
- [Background] Wang X, Perry AC. Metabolic and physiologic responses to video game play in 7- to 10-year-old boys. Arch Pediatr Adolesc Med. 2006 Apr;160(4):411-5. doi: 10.1001/archpedi.160.4.411. PMID 16585487
- [Background] Segal KR, Dietz WH. Physiologic responses to playing a video game. Am J Dis Child. 1991 Sep;145(9):1034-6. doi: 10.1001/archpedi.1991.02160090086030. PMID 1877563
- [Background] Ni Mhurchu C, Maddison R, Jiang Y, Jull A, Prapavessis H, Rodgers A. Couch potatoes to jumping beans: a pilot study of the effect of active video games on physical activity in children. Int J Behav Nutr Phys Act. 2008 Feb 7;5:8. doi: 10.1186/1479-5868-5-8. PMID 18257911
- [Background] Maddison R, Mhurchu CN, Jull A, Jiang Y, Prapavessis H, Rodgers A. Energy expended playing video console games: an opportunity to increase children's physical activity? Pediatr Exerc Sci. 2007 Aug;19(3):334-43. doi: 10.1123/pes.19.3.334. PMID 18019591
- [Background] Chin A Paw MJ, Jacobs WM, Vaessen EP, Titze S, van Mechelen W. The motivation of children to play an active video game. J Sci Med Sport. 2008 Apr;11(2):163-6. doi: 10.1016/j.jsams.2007.06.001. Epub 2007 Aug 13. PMID 17706461
- [Background] McDougall J DM. <br />Children, video games and physical activity. an exploratory study. Int J on Disability and Human Development. 2008;7(1):89-94.
- [Background] Spear BA, Barlow SE, Ervin C, Ludwig DS, Saelens BE, Schetzina KE, Taveras EM. Recommendations for treatment of child and adolescent overweight and obesity. Pediatrics. 2007 Dec;120 Suppl 4:S254-88. doi: 10.1542/peds.2007-2329F. PMID 18055654
- [Background] Whitlock EP, O'Connor EA, Williams SB, Beil TL, Lutz KW. Effectiveness of weight management interventions in children: a targeted systematic review for the USPSTF. Pediatrics. 2010 Feb;125(2):e396-418. doi: 10.1542/peds.2009-1955. Epub 2010 Jan 18. PMID 20083531
- [Background] Franklin J, Denyer G, Steinbeck KS, Caterson ID, Hill AJ. Obesity and risk of low self-esteem: a statewide survey of Australian children. Pediatrics. 2006 Dec;118(6):2481-7. doi: 10.1542/peds.2006-0511. PMID 17142534
- [Background] Cohen RY, Felix MR, Brownell KD. The role of parents and older peers in school-based cardiovascular prevention programs: implications for program development. Health Educ Q. 1989 Summer;16(2):245-53. doi: 10.1177/109019818901600208. PMID 2732066
- [Background] Ebbeling CB, Feldman HA, Osganian SK, Chomitz VR, Ellenbogen SJ, Ludwig DS. Effects of decreasing sugar-sweetened beverage consumption on body weight in adolescents: a randomized, controlled pilot study. Pediatrics. 2006 Mar;117(3):673-80. doi: 10.1542/peds.2005-0983. PMID 16510646
- [Background] Epstein LH, Valoski A, Wing RR, McCurley J. Ten-year outcomes of behavioral family-based treatment for childhood obesity. Health Psychol. 1994 Sep;13(5):373-83. doi: 10.1037//0278-6133.13.5.373. PMID 7805631
- [Background] Johnson G, Kent G, Leather J. Strengthening the parent-child relationship: a review of family interventions and their use in medical settings. Child Care Health Dev. 2005 Jan;31(1):25-32. doi: 10.1111/j.1365-2214.2005.00446.x. PMID 15658963
- [Background] Eklund RC, Whitehead JR, Welk GJ. Validity of the children and youth physical self-perception profile: a confirmatory factor analysis. Res Q Exerc Sport. 1997 Sep;68(3):249-56. doi: 10.1080/02701367.1997.10608004. No abstract available. PMID 9294879
- [Background] Whitehead JR. A study of children's physical self-perception using an adapted physical self-perception questionnaire. Pediatr Exercise Science. 1995(7):132-151.
- [Background] Block G, Hartman AM, Naughton D. A reduced dietary questionnaire: development and validation. Epidemiology. 1990 Jan;1(1):58-64. doi: 10.1097/00001648-199001000-00013. PMID 2081241
- [Background] Kamath CC, Vickers KS, Ehrlich A, McGovern L, Johnson J, Singhal V, Paulo R, Hettinger A, Erwin PJ, Montori VM. Clinical review: behavioral interventions to prevent childhood obesity: a systematic review and metaanalyses of randomized trials. J Clin Endocrinol Metab. 2008 Dec;93(12):4606-15. doi: 10.1210/jc.2006-2411. Epub 2008 Sep 9. PMID 18782880
- [Background] Epstein LH, Robinson JL, Temple JL, Roemmich JN, Marusewski A, Nadbrzuch R. Sensitization and habituation of motivated behavior in overweight and non-overweight children. Learn Motiv. 2008 Aug;39(3):243-255. doi: 10.1016/j.lmot.2008.03.001. PMID 19649135
- [Background] Proctor MH, Moore LL, Gao D, Cupples LA, Bradlee ML, Hood MY, Ellison RC. Television viewing and change in body fat from preschool to early adolescence: The Framingham Children's Study. Int J Obes Relat Metab Disord. 2003 Jul;27(7):827-33. doi: 10.1038/sj.ijo.0802294. PMID 12821969
- [Background] DeMattia L, Lemont L, Meurer L. Do interventions to limit sedentary behaviours change behaviour and reduce childhood obesity? A critical review of the literature. Obes Rev. 2007 Jan;8(1):69-81. doi: 10.1111/j.1467-789X.2006.00259.x. PMID 17212797
- [Background] Saunders TJ, Tremblay MS, Mathieu ME, Henderson M, O'Loughlin J, Tremblay A, Chaput JP; QUALITY cohort research group. Associations of sedentary behavior, sedentary bouts and breaks in sedentary time with cardiometabolic risk in children with a family history of obesity. PLoS One. 2013 Nov 20;8(11):e79143. doi: 10.1371/journal.pone.0079143. eCollection 2013. PMID 24278117
- [Background] Simons M, Bernaards C, Slinger J. Active gaming in Dutch adolescents: a descriptive study. Int J Behav Nutr Phys Act. 2012 Oct 2;9:118. doi: 10.1186/1479-5868-9-118. PMID 23031076
- [Background] Peng W, Crouse J. Playing in parallel: the effects of multiplayer modes in active video game on motivation and physical exertion. Cyberpsychol Behav Soc Netw. 2013 Jun;16(6):423-7. doi: 10.1089/cyber.2012.0384. Epub 2013 Mar 19. PMID 23509986
- [Background] Smallwood SR, Morris MM, Fallows SJ, Buckley JP. Are active video games useful in increasing physical activity and addressing obesity in children?--Reply. JAMA Pediatr. 2013 Jul;167(7):678. doi: 10.1001/jamapediatrics.2013.2421. No abstract available. PMID 23817856
- [Background] Baranowski T, Abdelsamad D, Baranowski J, O'Connor TM, Thompson D, Barnett A, Cerin E, Chen TA. Impact of an active video game on healthy children's physical activity. Pediatrics. 2012 Mar;129(3):e636-42. doi: 10.1542/peds.2011-2050. Epub 2012 Feb 27. PMID 22371457
- [Background] Lyons EJ, Tate DF, Ward DS, Wang X. Energy intake and expenditure during sedentary screen time and motion-controlled video gaming. Am J Clin Nutr. 2012 Aug;96(2):234-9. doi: 10.3945/ajcn.111.028423. Epub 2012 Jul 3. PMID 22760571
- [Background] Chaput JP, LeBlanc AG, Goldfield GS, Tremblay MS. Are active video games useful in increasing physical activity and addressing obesity in children? JAMA Pediatr. 2013 Jul;167(7):677-8. doi: 10.1001/jamapediatrics.2013.2424. No abstract available. PMID 23817855
- [Background] Barnett A, Cerin E, Baranowski T. Active video games for youth: a systematic review. J Phys Act Health. 2011 Jul;8(5):724-37. doi: 10.1123/jpah.8.5.724. PMID 21734319
- [Background] Biddiss E, Irwin J. Active video games to promote physical activity in children and youth: a systematic review. Arch Pediatr Adolesc Med. 2010 Jul;164(7):664-72. doi: 10.1001/archpediatrics.2010.104. PMID 20603468
- [Background] Gao Z, Hannan P, Xiang P, Stodden DF, Valdez VE. Video game-based exercise, Latino children's physical health, and academic achievement. Am J Prev Med. 2013 Mar;44(3 Suppl 3):S240-6. doi: 10.1016/j.amepre.2012.11.023. PMID 23415189
- [Background] Maddison R, Foley L, Ni Mhurchu C, Jiang Y, Jull A, Prapavessis H, Hohepa M, Rodgers A. Effects of active video games on body composition: a randomized controlled trial. Am J Clin Nutr. 2011 Jul;94(1):156-63. doi: 10.3945/ajcn.110.009142. Epub 2011 May 11. PMID 21562081
- [Background] Trost SG, Sundal D, Foster GD, Lent MR, Vojta D. Effects of a pediatric weight management program with and without active video games a randomized trial. JAMA Pediatr. 2014 May;168(5):407-13. doi: 10.1001/jamapediatrics.2013.3436. PMID 24589566
- [Background] Quinn M. Introduction of active video gaming into the middle school curriculum as a school-based childhood obesity intervention. J Pediatr Health Care. 2013 Jan;27(1):3-12. doi: 10.1016/j.pedhc.2011.03.011. Epub 2011 May 14. PMID 23237611
- [Background] Christison A, Khan HA. Exergaming for health: a community-based pediatric weight management program using active video gaming. Clin Pediatr (Phila). 2012 Apr;51(4):382-8. doi: 10.1177/0009922811429480. Epub 2011 Dec 8. PMID 22157430
- [Background] Guy S, Ratzki-Leewing A, Gwadry-Sridhar F. Moving beyond the stigma: systematic review of video games and their potential to combat obesity. Int J Hypertens. 2011;2011:179124. doi: 10.4061/2011/179124. Epub 2011 Mar 31. PMID 21629863
- [Background] Robertson W, Stewart-Brown S, Stallard N, Petrou S, Griffiths F, Thorogood M, Simkiss D, Lang R, Reddington K, Poole F, Rye G, Khan KA, Hamborg T, Kirby J. Evaluation of the effectiveness and cost-effectiveness of Families for Health V2 for the treatment of childhood obesity: study protocol for a randomized controlled trial. Trials. 2013 Mar 20;14:81. doi: 10.1186/1745-6215-14-81. PMID 23514100
- [Background] Okely AD, Collins CE, Morgan PJ, Jones RA, Warren JM, Cliff DP, Burrows TL, Colyvas K, Steele JR, Baur LA. Multi-site randomized controlled trial of a child-centered physical activity program, a parent-centered dietary-modification program, or both in overweight children: the HIKCUPS study. J Pediatr. 2010 Sep;157(3):388-94, 394.e1. doi: 10.1016/j.jpeds.2010.03.028. Epub 2010 May 6. PMID 20447648
- [Background] Baranowski T, Baranowski J, Thompson D, Buday R, Jago R, Griffith MJ, Islam N, Nguyen N, Watson KB. Video game play, child diet, and physical activity behavior change a randomized clinical trial. Am J Prev Med. 2011 Jan;40(1):33-8. doi: 10.1016/j.amepre.2010.09.029. PMID 21146765
- [Background] Davis MM, Gance-Cleveland B, Hassink S, Johnson R, Paradis G, Resnicow K. Recommendations for prevention of childhood obesity. Pediatrics. 2007 Dec;120 Suppl 4:S229-53. doi: 10.1542/peds.2007-2329E. PMID 18055653
- [Background] Mahar MT, Guerieri AM, Hanna MS, Kemble CD. Estimation of aerobic fitness from 20-m multistage shuttle run test performance. Am J Prev Med. 2011 Oct;41(4 Suppl 2):S117-23. doi: 10.1016/j.amepre.2011.07.008. PMID 21961611
- [Background] McNamara E, Hudson Z, Taylor SJ. Measuring activity levels of young people: the validity of pedometers. Br Med Bull. 2010;95:121-37. doi: 10.1093/bmb/ldq016. Epub 2010 Jun 18. PMID 20562207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Obese and overweight children (BMI ≥85th percentile) ages 8 through 12 years were referred to the program from their primary care practices or self-referred through advertisements distributed by the local park district and a community organization.
Pre-assignment Details: Participants with medical, developmental or psychiatric diagnoses which precluded participation in the curriculum or those taking medication that could significantly affect weight were excluded. Eighty-four subjects, mean age 10.1 years (SD 1.3 years), participated in the study from April 2011 through September 2013.
Groups:
- Exergaming and Didactic Health Teaching: Participation of child and parent/guardian in 6 months of weight management programming consisting of exergaming combined with didactic teaching.
  Exergaming and Didactic health teaching: 6 months of weight management programming consisting of 10 weekly 2- hour sessions:1 hour of exergaming and 1 hour of didactic classes teaching behavioral and dietary curricula. Followed by monthly 1-hour maintenance didactic teaching for the remainder of the 6 month period.
  n = 60 (71%) enrolled within 6 cohorts over the study period from April 2011 to September 2013.
- Didactic Health Teaching: Participation of child and parent/guardian in 6 months of weight management programming consisting only of didactic teaching.
  Didactic health teaching: 6 months of weight management programming consisting of 10 weekly 1-hour sessions of didactic classes teaching behavioral and dietary curricula. Followed by monthly 1-hour didactic health teaching sessions for the remainder of the 6 month period.
  n = 24 (29%) enrolled within 6 cohorts during the study period from April 2011 to September 2013
Period: Cohort 1
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Started | 14 | 4
Completed | 9 | 1
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Cohort 2
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Started | 14 | 10
Completed | 10 | 7
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 3
Period: Cohort 3
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Started | 12 | 0 (Enrollment too low to have control group. All subjects in this cohort received intervention.)
Completed | 7 | 0
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0
Period: Cohort 4
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Started | 6 | 0 (Enrollment too low to have control group. All subjects in this cohort received intervention.)
Completed | 4 | 0
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Cohort 5
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Started | 10 | 5
Completed | 4 | 1
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2
Period: Cohort 6
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Started | 4 | 5
Completed | 1 | 4
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: The subjects were enrolled sequentially and randomized 2:1 into two arms: the intervention group receiving both didactic and exergaming physical activity curriculum and the control group, who received didactic curriculum only. The control group were offered participation in the exergaming activities 6 months after randomization.
Groups:
- Exergaming and Didactic Health Teaching: Participation of child and parent/guardian in 6 months of weight management programming consisting of exergaming combined with didactic teaching.
  Exergaming and Didactic health teaching: 6 months of weight management programming consisting of 10 weekly 2- hour sessions:1 hour of exergaming and 1 hour of didactic classes teaching behavioral and dietary curricula. Followed by monthly 1-hour maintenance didactic teaching for the remainder of the 6 month period.
- Didactic Health Teaching: Participation of child and parent/guardian in 6 months of weight management programming consisting only of didactic teaching.
  Didactic health teaching: 6 months of weight management programming consisting of 10 weekly 1-hour sessions of didactic classes teaching behavioral and dietary curricula. Followed by monthly 1-hour didactic health teaching sessions for the remainder of the 6 month period.
- Total: Total of all reporting groups
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching | Total
Number analyzed (Participants) | 60 | 24 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] — Obese and overweight children (BMI greater than or equal to 85th percentile) ages 8 years through 12 years were enrolled.
  years | 10.0 (1.2) | 10.1 (1.1) | 10.1 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 12 | 49
  Male | 23 | 12 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 6 | 22
  White | 39 | 14 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline BMI z-score [Mean (Full Range); unit: z-score] | 2.2 [1.43 to 2.86] | 2.2 [1.27 to 2.96] | 2.2 [1.27 to 2.96]

OUTCOME MEASURES:

1. Primary Outcome: BMI Z-score Change
Description: All subjects were asked to dress in light athletic clothing and have their weight and height measured at baseline (the first group session) and at 6 months. Research assistants were trained using guidelines from the National Health and Nutrition Examination Survey (NHANES) Anthropometry Procedures Manual and demonstrated accurate measures on 3 separate children. The Seca 217 portable stadiometer was used for all height measurements and the HealthOMeter 844 KL scale was used for all weight measurements. BMI z-scores were calculated using software available from the Children's Hospital of Philadelphia Research Institute (http://stokes.chop.edu/web/zcore).
Time Frame: Change from baseline at 6 months
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 35 | 13
z-score | -0.057 (0.118) | 0.005 (0.0917)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.0967, t-test, 2 sided — We checked the distribution of bmiz changes between baseline and 6 months, and there is one subject from control group had bigger changes than others. After excluding this subject, the results are still similar with previous; Mean Difference (Net) = -0.0615, 95% CI 2-sided [-0.1344 to 0.0115]

2. Primary Outcome: BMI Z-score Change
Description: Measure was only taken on the subjects who participated in the Intervention group (exergaming combined with didactic teaching).
Time Frame: Change from baseline BMI z-score at 1 year
Population: Complete data was not available for all 35 subjects for this outcome measure. BMI z-score change from baseline to 1 year was only collected on 28 of the 35 participants.
Measure: Mean (95% Confidence Interval); unit: z-score
Groups:
- Exergaming and Didactic Health Teaching: Subjects remaining in the study at 1 year post start of participation in the exergaming combined with didactic health teaching sessions, 14 sessions over 6 month period, followed by 6 months of non-participation in group activity.
Arm/Group | Exergaming and Didactic Health Teaching
Number analyzed (Participants) | 28
z-score | -0.0775 [-0.1485 to -0.00652]
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching; Test type: Superiority or Other; p = 0.0335, t-test, 2 sided; Mean Difference (Net) = -0.0775, 95% CI 2-sided [-0.1485 to -0.00652]

3. Secondary Outcome: Waist Circumference Change
Time Frame: Change from baseline at 6 months
Population: Incomplete data available for analysis. Change in waist circumference from baseline to 6 month measurements was only collected on 34/35 of the Experimental group and 8/13 of the Active comparator group. The other participants did not show up for the 6 month measurements.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 34 | 8
cm | -0.50 (6.70) | -0.51 (5.12)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.991, t-test, 2 sided; Mean Difference (Net) = 0.0, 95% CI 2-sided [-5.2 to 5.1]

4. Secondary Outcome: Systolic Blood Pressure Change
Time Frame: Change from baseline Systolic BP at 6 months
Population: Incomplete data available for analysis. Blood pressure was taken and documented at baseline and at 6 months, however, not all participants were in attendance. Complete data was only available for 33/35 Experimental group participants and 12/13 from the Active comparator group. Available data was analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 33 | 12
mmHg | 1 (15) | 0 (15)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.851, t-test, 2 sided; Mean Difference (Net) = 1, 95% CI 2-sided [-9 to 11]

5. Secondary Outcome: Heart Rate Change From Baseline to 6 Months
Time Frame: Change from baseline at 6 months
Population: Missing Data: Heart rate measurements at baseline and at 6 months was only available for 33/35 Experimental group participants and 12/13 Active comparator group participants. Not all participants attended the 6 month measurement/data collection visit.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 33 | 12
beats per minute | -9.9 (13.77) | -7.0 (9.69)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.501, t-test, 2 sided; Mean Difference (Net) = -2.9, 95% CI 2-sided [-11.7 to 5.8]

6. Secondary Outcome: Shuttle Run Change in Number of Shuttle Runs
Description: The shuttle run was completed by participants at baseline (session 1) and at 6 months. The shuttle run is a standardized field assessment that requires participants to run 20 meters within sequentially shortened time frames of recorded beeps.
Time Frame: Change in number from baseline shuttle run at 6 months
Population: Missing Data: Shuttle run was completed by participants at baseline and at 6 months to document the change in number of runs. Not all participants attended the 6 month measurement visit, therefore, complete data was only available on 24/35 of the Experimental group and 13/13 of the Active comparator group. Available data was analyzed.
Measure: Mean (Standard Deviation); unit: number of runs
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 24 | 13
number of runs | 0.213 (0.4014) | -0.00085 (0.376)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.035, t-test, 2 sided; Mean Difference (Net) = 0.2971, 95% CI 2-sided [0.0224 to 0.5718]

7. Secondary Outcome: After School Screen Time as Reported on Questionnaire
Description: Change in after school screen time (reported out as fraction of 1 hour) will be measured by subject response on questionnaire taken at baseline and at 6 months for both groups. After school screen time was defined as the amount of time spent on any screen, on the average weekday afternoon/evening, including: watching television, computer use (laptop, desk top, tablet) or playing video games on the television or other hand held device.
Time Frame: Change from baseline at 6 months
Population: Missing Data: Survey data regarding "after school screen time" was collected from participants at baseline and again at 6 months. Not all participants completed both surveys, therefore, analysis for this outcome measure only included 28/35 participants from the Experimental group and 8/13 participants from the Active comparator group.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 28 | 8
hours | -0.7589 (3.068) | 0.188 (1.368)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.2207, t-test, 2 sided; Mean Difference (Net) = -0.9464, 95% CI 2-sided [-2.4954 to 0.6025]

8. Secondary Outcome: Saturday Screen Time as Assessed by Questionnaire
Description: Change in Saturday screen time (reported out as fraction of an hour) will be measured by subject response on questionnaire taken at baseline and at 6 months for both groups. Saturday screen time was defined as the amount of time spent on any screen, on an average Saturday, including: watching television, computer use (laptop, desk top, tablet) or playing video games on the television or other hand held device.
Time Frame: Change in hours from baseline at 6 months
Population: Missing Data: Survey data regarding "Saturday screen time" was collected from participants at baseline and again at 6 months. Not all participants completed both surveys, therefore, analysis for this outcome measure only included 28/35 participants from the Experimental group and 8/13 participants from the Active comparator group.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 28 | 8
hours | -1.4 (3.36) | -0.3438 (2.36)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.4164, t-test, 2 sided; Mean Difference (Net) = -1.0491, 95% CI 2-sided [-3.6407 to 1.5425]

9. Secondary Outcome: Activity Levels Measured by Pedometers (Weekly Steps)
Description: Activity will be measured by pedometers (number of steps) during week 1 and week 24 for both groups. Subjects used the Yamax 200 pedometer to count the steps they took over 1 weeks time.
Time Frame: Change from week 1 to week 24
Population: Missing data: Data was not available from all participants from pedometer use at both the 1 week and 24 week mark, therefore, this analysis only includes 13/35 participant data from the Experimental group and 10/13 participant data collected from the Active comparator group.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 13 | 10
steps | -6626 (21810) | -9059.5 (26688.91)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.812, t-test, 2 sided; Mean Difference (Net) = 2433.7, 95% CI 2-sided [-18579.7 to 23447.2]

10. Secondary Outcome: Self Perception as Assessed Using the Children and Youth Physical Self-Perception Profile (CY-PSPP): Physical Self-Worth Changes in Physical Self-worth
Description: CY-PSPP questionnaire was completed by participants in both groups at baseline and at 6 months. Change in the Physical Self-worth scores, which was 1 of 6 sub-domains, is analyzed. This sub-domain contains 6 questions with responses ranging from 1-4 for each question with 1 being the minimum and 4 being the maximum (best) score. The sub-domain score is then calculated as the mean of the 6 responses (minimum to maximum of 1 to 4).The change in score from baseline to 6 months was compared.
Time Frame: Change from baseline at 6 months
Population: Missing Data: The CY-PSPP questionnaire was not completed by all participants at both the baseline visit and the 6 month mark. Therefore this analysis only includes data for participants who completed the questionnaire at both times: 26/35 from the Experimental group and 7/13 from the Active Comparator group.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 26 | 7
scores on a scale | -0.218 (0.746) | -0.5 (0.385)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.3326, t-test, 2 sided; Mean Difference (Net) = 0.2837, 95% CI 2-sided [-0.3037 to 0.8711]

11. Secondary Outcome: Self Perception as Assessed Using the Children and Youth Physical Self-Perception Profile (CY-PSPP): Global Self-Worth Score
Description: CY-PSPP questionnaire was completed by participants in both groups at baseline and at 6 months. Change in the Global Self-worth scores, which was 1 of 6 sub-domains, is analyzed. This sub-domain contains 6 questions with responses ranging from 1-4 for each question with 1 being the minimum and 4 being the maximum (best) score. The sub-domain score is then calculated as the mean of the 6 responses (minimum to maximum of 1 to 4).The change in score from baseline to 6 months was compared.
Time Frame: Change from baseline to 6 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 26 | 7
scores on a scale | -0.238 (0.525) | -0.523 (0.53)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.1856, t-test, 2 sided; Mean Difference (Net) = 0.2995, 95% CI 2-sided [-0.2051 to 0.8041]

12. Secondary Outcome: Dietary Change:Total Calorie Intake (kcal/Day) (Block Alive FFQ)
Description: The Block Alive FFQ: administered at the start and at 6 months to all participants in both groups. FFQ inquires about typical dietary patterns over the previous six months. Total kcal/kg/day is then estimated based upon participant responses.
Time Frame: Change from baseline at 6 months
Population: Missing data: Not all participants completed this survey at both time points. 28/35 from the Experimental group had complete response and 10/13 from the Active comparator group had complete response. Analysis was completed on the available data.
Measure: Mean (Standard Deviation); unit: kcal/day
Groups:
- Exergaming and Didactic Health Teaching: Subjects attending exergaming/physical activity along with classroom structured nutrition/health education.
- Didactic Health Teaching: Subjects only receiving classroom structured nutrition/health education.
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 28 | 10
kcal/day | -292.92 (386.7) | -45 (358.5)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.0849, t-test, 2 sided; Mean Difference (Net) = -247.9, 95% CI 2-sided [-531.7 to 35.8686]

13. Secondary Outcome: Change in Dietary Intake: % Fat (Block Alive FFQ)
Description: The Block Alive FFQ: administered at the start and at 6 months to all participants in both groups. FFQ inquires about typical dietary patterns over the previous six months. Total %dietary fat intake per day is then estimated based upon participant responses.
Time Frame: Change from baseline at 6 months
Population: Missing data: Not all participants completed this survey at both time points. 28/35 from the Experimental group had complete response and 10/13 from the Active comparator group had complete response regarding the %fat in their daily diet. Analysis was completed on the available data.
Measure: Mean (Standard Deviation); unit: percentage of fat
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 28 | 10
percentage of fat | -1.25 (8.49) | 3.00 (7.09)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.176, t-test, 2 sided; Mean Difference (Net) = -4.2048, 95% CI 2-sided [-10.3835 to 1.9740]

14. Secondary Outcome: Change in Dietary Intake: % Carbohydrates (Block Alive FFQ)
Description: The Block Alive FFQ: administered at the start and at 6 months to all participants in both groups. FFQ inquires about typical dietary patterns over the previous six months. Total % dietary carbohydrates is then estimated based upon participant responses.
Time Frame: Change from baseline at 6 months
Population: Missing data: Not all participants completed this survey at both time points. 28/35 from the Experimental group had complete response and 10/13 from the Active comparator group had complete response regarding %carbohydrates in their daily diet. Analysis was completed on the available data.
Measure: Mean (Standard Deviation); unit: percentage of carbohydrates
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 28 | 10
percentage of carbohydrates | 2.10 (8.49) | -5.12 (7.95)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.0247, t-test, 2 sided; Mean Difference (Net) = 7.2151, 95% CI 2-sided [0.973 to 13.457]

15. Secondary Outcome: Change in Dietary Intake: Number of Vegetable Servings (Block Alive FFQ)
Description: The Block Alive FFQ: administered at the start and at 6 months to all participants in both groups. FFQ inquires about typical dietary patterns over the previous six months. Total number of vegetable servings per day is then estimated based upon participant responses.
Time Frame: Change from baseline at 6 months
Population: Missing data: Not all participants completed this survey at both time points. 25/35 from the Experimental group had complete response and 9/13 from the Active comparator group had complete response regarding daily vegetable intake. Analysis was completed on the available data.
Measure: Mean (Standard Deviation); unit: servings
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 25 | 9
servings | 0.0078 (0.7755) | 0.8248 (2.06)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.2764, t-test, 2 sided; Mean Difference (Net) = -0.8169, 95% CI 2-sided [-2.4147 to 0.7808]

16. Secondary Outcome: Change in Dietary Intake: Number of Fruit Servings (Block Alive FFQ)
Description: The Block Alive FFQ: administered at the start and at 6 months to all participants in both groups. FFQ inquires about typical dietary patterns over the previous six months. Total number of fruit servings per day is then estimated based upon participant responses.
Time Frame: Change from baseline at 6 months
Population: Missing data: Not all participants completed this survey at both time points. 25/35 from the Experimental group had complete response and 9/13 from the Active comparator group had complete response regarding daily fruit intake. Analysis was completed on the available data.
Measure: Mean (Standard Deviation); unit: Servings
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 25 | 9
Servings | -0.13255 (0.523) | 0.663 (0.64)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.0008, t-test, 2 sided; Mean Difference (Net) = -0.7958, 95% CI 2-sided [-1.2350 to -0.3566]

17. Secondary Outcome: Change in Dietary Intake: Number of Sugar Sweetened Beverages (Block Alive FFQ)
Description: The Block Alive FFQ: administered at the start and at 6 months to all participants in both groups. FFQ inquires about typical dietary patterns over the previous six months. Total number of sugar sweetened beverages per day is then estimated based upon participant responses.
Time Frame: Change from baseline at 6 months
Population: Missing data: Not all participants completed this survey at both time points. 27/35 from the Experimental group had complete response and 10/13 from the Active comparator group had complete response regarding sugar sweetened beverage daily intake. Analysis was completed on the available data.
Measure: Mean (Standard Deviation); unit: servings
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Number analyzed (Participants) | 27 | 10
servings | -2.572 (8.402) | -3.2374 (2.44)
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching vs Didactic Health Teaching; Test type: Superiority or Other; p = 0.6974, t-test, 2 sided; Mean Difference (Net) = 0.7024, 95% CI 2-sided [-2.9377 to 4.3425]

18. Secondary Outcome: Exergaming Program Component Influence on Attendance
Description: The experimental group will answer a questionnaire at the end of the 6 month study period, measuring the importance of specific components of the curriculum and motivators which influenced enrollment and compliance with participation. Of interest is measuring the influence of the exergaming curriculum as compared to these other factors. This is a 16-item, 3-point Likert-scale (1 = least important and 3 = most important) questionnaire created specifically for this study. Results were reported based on % of participants rating "3" ,most important, for each curriculum component.
Time Frame: 6 months
Measure: Number; unit: percentage of subjects
Groups:
- Exergaming and Didactic Health Teaching: Intervention group subjects (exergaming combined with didactic nutrition teaching) with continued participation at 6 months completed this questionnaire regarding attitudes/perceptions towards participation.
Arm/Group | Exergaming and Didactic Health Teaching
Number analyzed (Participants) | 35
percentage of subjects | 71

19. Secondary Outcome: Waist Circumference Change
Time Frame: Change from 6 month waist circumference at 1 year
Population: One year data was only collected for the participants assigned to the "Exergaming and Didactic Health Teaching" group. Only 25/35 participants had waist measurements collected at both 6 months and 1 year. Available data was analyzed.
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Exergaming and Didactic Health Teaching
Number analyzed (Participants) | 25
cm | 1.52 [-0.9278 to 3.9678]
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching; Test type: Superiority or Other; p = 0.2122, t-test, 2 sided

20. Secondary Outcome: Systolic Blood Pressure Change
Time Frame: Change from 6 month Systolic BP at 1 year
Population: One year data was only collected for the participants assigned to the "Exergaming and Didactic Health Teaching" group. Systolic blood pressure was only documented at 6 months and 1 year for 27/35 of the participants. Available data is what was analyzed.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Exergaming and Didactic Health Teaching
Number analyzed (Participants) | 27
mmHg | 3.5185 [-1.0625 to 8.0996]
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching; Test type: Superiority or Other; p = 0.1265, t-test, 2 sided; Mean Difference (Net) = 3.61, 95% CI 2-sided [-1.15 to 8.33]

21. Secondary Outcome: Heart Rate Change
Time Frame: Change from 6 month Heart rate at 1 year
Population: One year data was only collected for the participants assigned to the "Exergaming and Didactic Health Teaching" group. Heart rate data was collected at 6 month and 1 year for 27/35 of the participants. Available data was analyzed.
Measure: Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | Exergaming and Didactic Health Teaching
Number analyzed (Participants) | 27
beats per minute | 2.7407 [-3.3961 to 8.8776]
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching; Test type: Superiority or Other; p = 0.3671, t-test, 2 sided

22. Secondary Outcome: Shuttle Run Change in Number of Shuttle Runs
Description: The shuttle run was completed again by participants in the Experimental group at 1 year. The shuttle run is a standardized field assessment that requires participants to run 20 meters within sequentially shortened time frames of recorded beeps.
Time Frame: Change in number from 6 month shuttle run at 1 year
Population: One year data was only collected for the participants assigned to the "Exergaming and Didactic Health Teaching" group. Shuttle run was completed by 20/35 participants in the Experimental group at both 6 months and 1 year. Available data was analyzed.
Measure: Mean (95% Confidence Interval); unit: number of runs
Arm/Group | Exergaming and Didactic Health Teaching
Number analyzed (Participants) | 20
number of runs | 0.10 [-0.1968 to 0.3968]
Statistical Analysis 1: Comparison: Exergaming and Didactic Health Teaching; Test type: Superiority or Other; p = 0.4892, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse Event data collected throughout the length of the study for all participants (12 month participation period).
Arm/Group | Exergaming and Didactic Health Teaching | Didactic Health Teaching
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/24
Other Adverse Events (participants affected / at risk) | 0/60 | 0/24

LIMITATIONS AND CAVEATS:
Limitations: incomplete data collection (baseline & follow-up), those lost to follow-up may have been unwilling to continue because of weight gain, low enrollment numbers, and control subjects were offered intervention activities after 6 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No